CLINICAL TRIAL: NCT01047670
Title: Reposição de Esteróides em Crianças Com Choque Séptico
Brief Title: Septic Shock em Steroids
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unidade de Terapia Intensiva (Other)
Responsible Party: Pedro Celiny Ramos Garcia, Pontifícia Universidade Católica do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Esteroides725
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2008-03

CONDITIONS: Mechanical Ventilation; Mortality
Keywords: sepsis, shock, adrenal insufficiency, hydrocortisone, children, paediatric intensive care.; number of days free of vasoactive support in 7 days; days free of mechanical ventilation; PICU mortality; mortality among patient with inappropriate response to the ACTH test; baseline cortisol/ PIM2 correlation
MeSH Terms: conditions — Sepsis; Shock; Adrenal Insufficiency | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Hydrocortisone 6 mg/kg/day, 8 hourly, during 7 days or during the vasoactive drug infusion
  Interventions: Drug: Hydrocortisone
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone 6 mg/kg/day, 8 hourly, during 7 days or during the vasoactive drug infusion

SUMMARY:
Septic shock is a frequent reason for admission on pediatric intensive care units. Interventions which can change morbidity and mortality of septic shock patients are of great interest. Steroid replacement in adults with severe sepsis and septic shock have been extensively studied. It was recently demonstrated that low dose steroid (< 300mg/ day) used for more than 5 days was associated with decreased mortality and lower requirement of vasoactive support in the adult population that had a low response to the ACTH test. However, this was not confirmed in the latest results from the CORTICUS study. Use of low dose hydrocortisone, or any other steroid has not been studied in critically ill children. Mortality associated with sepsis in children has decreased in the last decade and currently it is close to 10%, making it difficult to power a study able to show reduced mortality. Taking into account the results from previous studies reporting the high incidence of adrenal failure and its association to worse outcome, we have designed a clinical trial to evaluate the effect of low dose hydrocortisone in children with septic shock: Cortisol Replacement in Children with Sepsis Study.

DETAILED DESCRIPTION:
Hypothesis Pediatric patients with septic shock have a high incidence of failure to respond to the ACTH test and would benefit of steroid replacement.

Design Randomized double-blind placebo controlled clinical trail. Outcome Primary: number of days free of vasoactive support after 7 days of septic shock diagnosis.

Methods

Study population:

All children admitted to PICU will be possible enrolled. Inclusion criteria will be (I) age between 1 month and 16 years; (II) septic shock according to the definitions of pediatric septic shock 2005; (III) inotrope requirement, as in dopamine > 5 mcg/kg/mim, dobutamine > 5 mcg/kg/min or any dose of noradrenaline or adrenaline after adequate fluid resuscitation. Exclusion criteria will be patients with (I) baseline disease associated to HPA axis dysfunction; (II) steroid use in the past 4 weeks; (III) previous use of etomidate; (IV) formal indication for steroids use, and (V) formal contraindication to steroid use.

Stratification criteria:

Patients will be stratified by age, gender, PRISM category, failure to respond to ACTH test, surgical patients, chronic patient, baseline cardiac and oncological disease and presence of ARDS.

Intervention:

Hydrocortisone 6 mg/kg/day, 8 hourly, during 7 days or during the vasoactive drug infusion. The control group will receive placebo.

Randomization:

Randomization will be carried through numbered envelopes, randomized prior to the study beginning, in blocks of 10, ratio 1:1.

Protocol:

Identical vials with hydrocortisone or placebo will be prepared in an industrial pharmacy and labeled using alphabetic letters (A, B, C, D) before the beginning of the study. Each vial of hydrocortisone will have 100 mg of hydrocortisone ponder to be diluted in 10 ml of normal saline 0.9% Each vial of placebo will content a innocuous ponder, also to be diluted in 10 ml of normal saline 0.9%. The drug and its referent letter (A, B, C, D) will be controlled by two lists, handed in by the pharmacist to the researchers inside closed envelopes before the beginning of the study. After enrollment and randomization, children joining the study will have baseline cortisol and ACTH measured. ACTH testes (1 mcg/ 1.75m2 and 250 mcg) will be performed, 4 hours apart. After this, patients will receive the study drug (either hydrocortisone or placebo), 0.2 ml/kg/ dose, 8 hourly. This will last the period the patient requires vasoactive support, or a maximum of 7 days. Daily routine blood results will be noted, as well as a further ACTH test on day 3 if the patient is still on vasoactive support. Demographic data will be collected on enrollment.

ELIGIBILITY:
Inclusion Criteria:

* (I) age between 1 month and 20 years;
* (II) septic shock according to the definitions of paediatric septic shock 2005; -(III) inotrope requirement, as in dopamine > 5 mcg/kg/mim, dobutamine > 5 mcg/kg/min or any dose of noradrenaline or adrenaline after adequate fluid resuscitation. -

Exclusion Criteria:

Exclusion criteria will be patients with

* (I) baseline disease associated to HPA axis dysfunction;
* (II) steroid use in the past 4 weeks;
* (III) previous use of etomidate; (IV) formal indication for steroids use, and
* (V) formal contraindication to steroid use.

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2008-05

PRIMARY OUTCOMES:
number of days free of vasoactive support after 7 days of septic shock diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul, Brazil